CLINICAL TRIAL: NCT01633827
Title: Combination Therapy for the Treatment of Obstructive Sleep Apnea
Brief Title: Combination Therapy to Treat Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Andrew Wellman, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BWH-2012P000956; 5R01HL102321-02 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-07-04 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Sugars; Hypnotics and Sedatives; Eszopiclone; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive both a sugar pill and room air during their overnight sleep studies
  Interventions: Drug: Placebo pill; Other: Room air
- Treatment (Active Comparator): Subjects will receive both Lunesta (eszopiclone) and medical grade oxygen during their overnight sleep studies
  Interventions: Drug: Sedative; Other: Oxygen

INTERVENTIONS:
Drug: Placebo pill — Subjects will receive a sugar pill (in combination with room air) during their placebo arm studies
  Other Names: sugar pill
  Arms: Placebo
Drug: Sedative — Subjects will receive eszopiclone (in combination with medical oxygen) during their treatment arm studies
  Other Names: Lunesta
  Arms: Treatment
Other: Room air — Subjects will receive room air (in combination with a sugar pill) during their placebo arm studies
  Arms: Placebo
Other: Oxygen — Subjects will receive medical grade oxygen (in combination with eszopiclone) during their treatment arm studies
  Arms: Treatment

SUMMARY:
In Obstructive sleep apnea (OSA), the upper airway closes over and over again during sleep. This leads to disrupted sleep (waking up during the night), daytime sleepiness, and an increased risk for developing high blood pressure. Currently, the best treatment for obstructive sleep apnea is sleeping with a mask that continuously blows air into the nose (i.e. Continuous positive airway pressure [CPAP] treatment). While CPAP treatment stops the upper airway from closing in most people, many people have difficulty sleeping with the mask in place and therefore do not use the CPAP treatment. This research study is being conducted to learn whether using a combination of therapies (i.e. a sedative and oxygen therapy) will improve OSA severity by altering some of the traits that are responsible for the disorder.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive collapse or 'obstruction' of the pharyngeal airway during sleep. These obstructions result in repetitive hypopneas/apneas and intermittent hypoxia/hypercapnia, as well as surges in sympathetic activity. Such processes disturb normal sleep and impair neurocognitive function, often resulting in excessive daytime sleepiness and decreased quality of life. Furthermore, OSA is associated with cardiovascular morbidity and mortality, making OSA a major health concern.

Current evidence suggests that OSA pathogenesis involves the interactions of at least four physiological traits comprising 1) the pharyngeal anatomy and its propensity towards collapse 2) the ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation), 3) the arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep) and 4) the stability of the ventilatory feedback loop (i.e. loop gain). Continuous positive airway pressure (CPAP) is the most common treatment for OSA but it is often poorly tolerated; only ~50% of patients diagnosed with OSA continue therapy beyond 3 months. Given this limitation, alternative approaches have been tested and have generally focused on the use of oral appliances, surgery, and more recently pharmacological agents.

However, these alternate therapies, when used alone as monotherapy, rarely abolish OSA completely. This is not that surprising given that these treatments focus primarily on correcting only one trait and ignore the fact that the pathogenesis of OSA is multi-factorial. Thus the investigators hypothesize that some patients could be treated without CPAP if more than one trait is targeted (i.e., the investigators take a multi-factorial treatment approach). Such a multi-factorial approach is not unusual in Medicine. Many disorders such as diabetes, asthma, hypertension, cancer and congestive heart failure are treated with more than one medication or modality. In our view, giving CPAP to all OSA patients is like treating every diabetic with insulin, or every asthmatic with oral steroids - these treatments, like CPAP, are poorly tolerated and ignore the complexity of the underlying biology.

The investigators recently published a technique that measures the four traits using repeated 'drops' in CPAP levels during sleep. Each trait is measured in a way that allows model-based predictions of the presence/absence of OSA. With this technique the investigators demonstrated in a small group of CPAP-treated OSA subjects that decreasing the sensitivity of the ventilatory feedback loop (i.e. reducing loop gain) by approximately 50% with either acetazolamide or oxygen reduces the apnea/hypopnea index (AHI) by half. Interestingly, our model allowed us to make the prediction that if, in addition to an agent that reduces loop gain, the investigators also gave a drug that increases the arousal threshold by at least 25%, then the investigators could potentially abolish OSA (rather than just reduce its severity by 50%). This is of great interest given that the investigators already have shown than eszopiclone increases the arousal threshold by approximately 30% and is associated with an improvement in the AHI. However, to date there has been no study examining the combination of an agent that reduces loop gain (i.e. oxygen) with one that increases the arousal threshold (i.e. eszopiclone) as a treatment for OSA.

To determine the effect of combination therapy on each of the four traits and how they contribute to our model prediction of OSA, as well as on apnea severity. Specifically the investigators will assess:

1. The physiological traits responsible for OSA:

   1. Pharyngeal anatomy and its propensity towards collapse
   2. The ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation)
   3. Arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep).
   4. Stability of the ventilatory control system feedback loop (i.e. loop gain)
2. The severity of OSA (apnea-hypopnea index (AHI), percent of time with unstable breathing, sleep quality)

STUDY DESIGN:

A single-blinded randomized control design will be used. Initially, participants will be randomized to either the treatment or placebo arm where they will have both a clinical and research polysomnography (PSG); these initial PSGs constitute what will be referred to as VISIT 1 (see outcome measures). The purpose of the clinical PSG is to determine the severity of OSA (i.e. AHI). The research PSG will measure the 4 physiological OSA traits.

During the treatment arm, in both PSGs (i.e. clinical and research) participants will be given eszopiclone (3mg by mouth) to take before bed and be placed on oxygen throughout the night. During the placebo arm, subjects will be given a placebo to take before bed and placed on room air while they sleep. Participants will then have at least a 1-week washout period and cross over to the other arm of the study whereby the clinical and research PSG will be repeated; these studies constitute what will be referred to asVISIT 2 (see outcome measures).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 79 years
* Documented OSA (AHI > 10 events/hr Non rapid eye movement sleep supine)
* If treated then, current CPAP use (>4 hrs CPAP/night for > 2 months)

Exclusion Criteria:

* Any uncontrolled medical condition
* Any other sleep disorder (Periodic leg movement syndrome, restless legs syndrome, insomnia, etc.)
* Use of medications known to affect sleep/arousal, breathing, or muscle physiology
* Allergy to lidocaine or Afrin
* Claustrophobia
* Alcohol consumption within 24 hours of PSG

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Wellman, MD, Principal Investigator — Brigham & Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Landry SA, Joosten SA, Sands SA, White DP, Malhotra A, Wellman A, Hamilton GS, Edwards BA. Response to a combination of oxygen and a hypnotic as treatment for obstructive sleep apnoea is predicted by a patient's therapeutic CPAP requirement. Respirology. 2017 Aug;22(6):1219-1224. doi: 10.1111/resp.13044. Epub 2017 Apr 13. PMID 28409851
- [Derived] Edwards BA, Sands SA, Owens RL, Eckert DJ, Landry S, White DP, Malhotra A, Wellman A. The Combination of Supplemental Oxygen and a Hypnotic Markedly Improves Obstructive Sleep Apnea in Patients with a Mild to Moderate Upper Airway Collapsibility. Sleep. 2016 Nov 1;39(11):1973-1983. doi: 10.5665/sleep.6226. PMID 27634790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a previous diagnosis of OSA (defined as an apnoea/hypopnoea index [AHI] >10/hr) were recruited from the sleep clinic and Brigham and Women's Hospital and the general community (Boston, MA). The first patient was recruited in September 2012 and the last patient enrolled in May 2014.
Groups:
- Placebo and Air First, Then Eszopiclone and Oxygen: Subjects will receive both a sugar pill and room air during two overnight sleep studies first and subsequently eszopiclone 3 mg with oxygen (FiO2 0.4) after a washout period of 1 week.
- Eszopiclone and Oxygen First, Then Placebo and Air: Subjects will receive both eszopiclone and medical grade oxygen (FIO2 0.4) during two overnight sleep studies, after a washout period of 1 week they will receive placebo and air during two overnight sleep studies
Period: First Intervention
Arm/Group | Placebo and Air First, Then Eszopiclone and Oxygen | Eszopiclone and Oxygen First, Then Placebo and Air
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Placebo and Air First, Then Eszopiclone and Oxygen | Eszopiclone and Oxygen First, Then Placebo and Air
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo and Air First, Then Eszopiclone and Oxygen | Eszopiclone and Oxygen First, Then Placebo and Air
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: During the placebo arm, one participant did not have OSA and another exhibited predominantly central sleep apnoea; both were excluded from the analysis.
Groups:
- Study Group: This study was a randomized cross-over design so each particiapnt enrolled underweent both placebo and treatment conditions.
  During the placebo arm, one participant did not have OSA and another exhibited predominantly central sleep apnea; both were excluded from the analysis. Subject demographics for the 20 remaining unselected patients are shown below.
Arm/Group | Study Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.8)
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Model Prediction of Absence/Presence of OSA: Ventilation That Causes an Arousal From Sleep (Varousal)
Description: Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual.
  In this table the investigators report the minimum ventilation that can be tolerated before an arousal from sleep (Varousal). It is calculated by slowly reducing the CPAP level from optimum to the minimum tolerable pressure. This trait is symbolized as Varousal (L/min)
Time Frame: Subjects will be assessed on day 1 (visit 1) and up to 1 month (visit 2)
Population: During the placebo arm, one participant did not have OSA and another exhibited predominantly central sleep apnea; both were excluded from the analysis. Subject results for the 20 remaining patients are reported here per intervention.
Measure: Mean (Standard Error); unit: L/min
Groups:
- Placebo Data: These result reports the minimum ventilation that can be tolerated before an arousal from sleep under placebo and room air administration
- Treatment Data: These result reports the minimum ventilation that can be tolerated before an arousal from sleep under the conditions of oxygen and a sedative.
Arm/Group | Placebo Data | Treatment Data
Number analyzed (Participants) | 20 | 20
L/min | 5.7 (0.3) | 5.2 (0.3)
Statistical Analysis 1: Comparison: Placebo Data vs Treatment Data; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.05

2. Primary Outcome: Model Prediction of Absence/Presence of OSA: Ventilatory Control Sensitivity (Loop Gain)
Description: Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual and predicts OSA presence/absence.
  In this table the investigators report the ventilatory control sensitivity value (Loop Gain). It is calculated dividing the increase in ventilatory drive by the steady state reduction in ventilation. The increase in ventilatory drive is measured as the ventilatory overshoot following a switch to optimal CPAP from the minimum tolerable CPAP. This trait is symbolized as steady state loop gain (LG, adimensional)
Time Frame: Subjects will be assessed on day 1 (visit 1) and up to 1 month (visit 2)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio, adimensional
Groups:
- Placebo Data: These results report the ventilatory control sensitivity (i.e., loop gain) during placebo and room air administration
- Treatment Data: These result report the ventilatory control sensitivity (i.e., loop gain) during eszopiclone and oxygen administration
Arm/Group | Placebo Data | Treatment Data
Number analyzed (Participants) | 20 | 20
ratio, adimensional | 3.3 (0.5) | 2.20 (0.25)
Statistical Analysis 1: Comparison: Placebo Data vs Treatment Data; Test type: Superiority or Other; p = 0.025, t-test, 2 sided; Mean Difference (Final Values) = 0.025

3. Primary Outcome: Model Prediction of Absence/Presence of OSA: Passive Collapsibility
Description: Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual and predicts OSA presence/absence.
  The passive collapsibility of the upper airway is quantified as the ventilation on no CPAP (atmospheric pressure) at the eupneic level of ventilatory drive when upper airway dilator muscles are relatively passive. This trait is symbolized as Vpassive (L/min)
Time Frame: Subjects will be assessed on day 1 (visit 1) and up to 1 month (visit 2)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/min
Groups:
- Placebo Data: These results represent the ventilation through a passive airway (when pharyngeal dilator muscles are not recruited) at atmospheric pressure and eupneic ventilatory drive during the administration of placebo and room air
- Treatment Data: These results represent the ventilation through a passive airway (when pharyngeal dilator muscles are not recruited) at atmospheric pressure and eupneic ventilatory drive during eszopiclone and oxygen administration
Arm/Group | Placebo Data | Treatment Data
Number analyzed (Participants) | 20 | 20
L/min | 1.40 (0.5) | 1.20 (0.41)
Statistical Analysis 1: Comparison: Placebo Data vs Treatment Data; Test type: Superiority or Other; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = 0.5

4. Primary Outcome: Model Prediction of Absence/Presence of OSA: Active Collapsibility (Vactive)
Description: Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual and predicts OSA presence/absence.
  Active collapsibility is the ventilation on no CPAP when upper airway muscle are maximally activated. It is calculated by slowing reducing CPAP from the optimal to the minimum tolerable level and rapidly dropping the CPAP to 0 for a few breaths. This trait is symbolized as Vactive (L/min)
Time Frame: Subjects will be assessed on day 1 (visit 1) and up to 1 month (visit 2)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: L/min
Groups:
- Placebo Data: These results represent the ventilation through a active airway (when pharyngeal dilator muscles maximally recruited) at atmospheric pressure during the administration of placebo and room air
- Treatment Data: These results represent the ventilation through a active airway (when pharyngeal dilator muscles maximally recruited) at atmospheric pressure during eszopiclone and oxygen administration
Arm/Group | Placebo Data | Treatment Data
Number analyzed (Participants) | 20 | 20
L/min | 4.4 (0.5) | 4 (0.45)
Statistical Analysis 1: Comparison: Placebo Data vs Treatment Data; Test type: Superiority or Other; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = 0.5

5. Secondary Outcome: Apnea-Hypopnea Index
Description: The Apnea-Hypopnea Index (AHI) is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow).
Time Frame: Subjects will be assessed on day 1 (visit 1) and up to 1 month (visit 2)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events/hr
Groups:
- Placebo Data: This result reports the AHI under the conditions of room air and a placebo tablet.
- Treatment Data: This result reports the AHI under the conditions of oxygen and eszopiclone
Arm/Group | Placebo Data | Treatment Data
Number analyzed (Participants) | 20 | 20
events/hr | 51.9 (6.2) | 29.5 (5.3)
Statistical Analysis 1: Comparison: Placebo Data vs Treatment Data; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 0.001

ADVERSE EVENTS:
Groups:
- Study Group: This study was a randomized cross-over design so each particiapnt enrolled underweent both placebo and treatment conditions
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
The overall limitation is that we have only assessed the impact of combination therapy on one night. Thus, longitudinal studies will be needed to determine if the treatments remain effective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No